CLINICAL TRIAL: NCT03754582
Title: A Multicenter, Uncontrolled, Open-label Study to Evaluate the Safety and Tolerability of Intravenous Perampanel as Substitute for Oral Tablet in Subjects With Partial Onset Seizures (Including Secondarily Generalized Seizures) or Primary Generalized Tonic-clonic Seizures
Brief Title: A Study of Intravenous Perampanel in Japanese Participants With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-J081-240
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-11

CONDITIONS: Epilepsy; Seizures
Keywords: Partial Onset Seizures; Secondarily Generalized Seizures; Primary Generalized Tonic-Clonic Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perampanel (Experimental): Participants with POS with or without secondarily generalized seizures or PGTC seizures will receive perampanel 8 to 12 milligram (mg), tablets, orally, once daily for 28 days (Day -28 to Day -1) in Pretreatment Phase and followed by 8 to 12 mg dose of perampanel as intravenous infusion for 30 minutes, once daily from Day 1 to Day 4 in Treatment Phase, and then again 8 to 12 mg, tablets, orally, once daily from Day 5 to Day 11 in Follow-up Phase as an adjunctive therapy, along with 1 to a maximum of 3 marketed concomitant antiepileptic drugs (AEDs).
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Oral tablets.
  Other Names: E2007
Drug: Perampanel — Intravenous infusion.
  Other Names: E2007

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of perampanel administered as a 30-minute intravenous infusion after switching from oral tablets (8 to 12 milligrams per day [mg/day]) as an adjunctive therapy in participants with epilepsy with partial onset seizures (POS) (including secondarily generalized seizures) or primary generalized tonic-clonic (PGTC) seizures.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of epilepsy with POS (including secondarily generalized seizures) or PGTC seizures according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures (1981).
2. Receiving a stable dose regimen of oral perampanel.
3. Receiving a concomitant stable dose regimen of marketed AEDs. No change of dosing regimen for concomitant AEDs is planned during the intravenous Treatment and Follow-up Phases.
4. Considered reliable and willing to be available for the study period by the investigator, and are able to record seizures and report AEs by themselves or have a caregiver who can record seizures and report AEs for them.

Exclusion Criteria:

1. A history of drug or alcohol dependency or abuse.
2. A history of status epilepticus.
3. Unsuitable for venipuncture and intravenous administration.
4. Requires medical intervention due to safety issues related to concomitant administration of AEDs.
5. A history of suicidal ideation/attempt.
6. Clinical symptoms or imaging suggest progressive central nervous system (CNS) abnormality, disorder, or brain tumor.
7. Current evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigators could affect the participant's safety, interfere with the study assessments or need prohibited medications as specified in the study protocol.
8. Clinically significant abnormal laboratory values.
9. Females of childbearing potential who:

   * In the Pretreatment Phase, are breastfeeding or pregnant (as documented by a positive beta-human chorionic gonadotropin [β-hCG] test).
   * Within 28 days before Visit 1, did not use a highly effective method of contraception, which includes any of the following:

     * total abstinence (if it is their preferred and usual lifestyle).
     * an intrauterine device (IUD) or intrauterine hormone-releasing system (IUS).
     * a contraceptive implant.
     * an oral contraceptive (with additional barrier method). (Participant must be on a stable dose of the same oral contraceptive product for at least 28 days before Day 1 of the Treatment Phase and throughout the entire study period, and for 28 days after the last dose of study drug).
     * have a vasectomized partner with confirmed azoospermia.
     * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after the last dose of study drug.
10. Participation in a study involving administration of an investigational drug or device within 28 days before Visit 1, or within approximately 5 half-lives of the previous investigational compound, whichever is longer.
11. A prolonged QT interval corrected using Fridericia's formula (QTcF) interval (greater than [>] 450 millisecond [ms]) as demonstrated by a repeated ECG.
12. A vagus nerve stimulation (VNS) implanted.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (13):
  - Eisai trial site 5, Kurume, Fukuoka
  - Eisai trial site 12, Sapporo, Hokkaido
  - Eisai trial site 9, Ōmura, Nagasaki
  - Eisai trial site 7, Sayama, Osaka
  - Eisai trial site 2, Asaka, Saitama
  - Eisai trial site 13, Hamamatsu, Shizuoka
  - Eisai trial site 8, Kodaira, Tokyo
  - Eisai trial site 10, Hiroshima
  - Eisai trial site 6, Kagoshima
  - Eisai trial site 1, Niigata
  - Eisai trial site 11, Okayama
  - Eisai trial site 3, Shizuoka
  - Eisai trial site 4, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 13 investigative sites in Japan from 27 November 2018 to 10 December 2019.
Pre-assignment Details: A total of 27 participants were consented, of which 6 were screen failures and 21 were enrolled and received the study treatment.
Groups:
- Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day: Participants with partial onset-seizures (POS) with or without secondarily generalized seizures or primary generalized tonic clonic (PGTC) seizures received perampanel 8 milligram (mg) up to 12 mg (stable-dosage), tablets, orally, once daily for 28 days (Day -28 to Day -1) as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant antiepileptic drugs (AEDs). Eligible participants who completed Pretreatment Phase entered in Treatment Phase.
- Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures were hospitalized and received perampanel 8 mg up to 12 mg (stable-dosage) equivalent to the oral dose, as intravenous infusion for 30 minutes, once daily on Day 1 to Day 4 as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs. Eligible participants who completed Treatment Phase entered Follow-up Phase.
- Follow-up Phase: Oral Perampanel 8 to 12 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures received perampanel 8 mg up to 12 mg (stable-dosage), tablets, orally, once daily on Day 5 to Day 11 (Follow-up Visit) as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs.
Period: Pretreatment Phase
Arm/Group | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Started | 21 | 0 | 0
Completed | 21 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Phase
Arm/Group | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Started | 0 | 21 | 0
Completed | 0 | 20 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Follow-up Phase
Arm/Group | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Started | 0 | 0 | 21 (1 participant who discontinued in Treatment Phase was assessed at Follow-up Visit.)
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Perampanel 8 to 12 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures received maintenance dose of perampanel 8 to 12 mg, tablets, orally, once daily for 28 days (Day -28 to Day -1) in Pretreatment Phase followed by 8 to 12 mg maintenance dose of perampanel equivalent to the oral dose, as intravenous infusion for 30 minutes, once daily from Day 1 to Day 4 in Treatment Phase, and then 8 to 12 mg maintenance dose of perampanel, tablets, orally, once daily from Day 5 to Day 11 (Follow-up Visit) in Follow-up Phase as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs.
Arm/Group | Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE was defined as any untoward medical occurrence that at any dose: Resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect.
Time Frame: Up to 60 days (Pretreatment Phase: up to 28 days, Treatment Phase: up to 4 days, Follow-up Phase: up to 28 days after last dose)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures received perampanel 8 mg up to 12 mg (stable-dosage), tablets, orally, once daily for 28 days (Day -28 to Day -1) as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs. Eligible participants who completed Pretreatment Phase entered in Treatment Phase.
Arm/Group | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21 | 21 | 21
Participants | 0 | 1 | 2

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product, any new disease or exacerbation of an existing disease, any deterioration in nonprotocol-required measurements of a laboratory value or other clinical test that resulted in symptoms, a change in treatment, or discontinuation of study drug, recurrence of an intermittent medical condition not present pretreatment, an abnormal laboratory test result was considered an AE if the identified laboratory abnormality led to any type of intervention, withdrawal of study drug, or withholding of study drug, whether prescribed in the protocol or not.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21 | 21 | 21
Participants | 3 | 15 | 6

3. Primary Outcome: Number of Participants With Markedly Abnormal Clinical Laboratory Parameter Values During Treatment and Follow-up Phase
Time Frame: Up to Day 11 (Treatment Phase: at Day 4, Follow-up Phase: up to 7 days after last dose)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21 | 21
Participants
  Triglycerides: Markedly Abnormal High | 1 | 0
  Urate: Markedly Abnormal High | 0 | 1

4. Primary Outcome: Number of Participants With Abnormal Vital Sign Values During Treatment and Follow-up Phase
Time Frame: Up to 11 days (Treatment Phase: up to 4 days, Follow-up Phase: up to 7 days after the last dose)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21 | 21
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Body Weight During Treatment and Follow-up Phase
Time Frame: Up to 11 days (Treatment Phase: up to 4 days, Follow-up Phase: up to 7 days after the last dose)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21 | 21
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Markedly Abnormal Electrocardiogram (ECG) Value During Treatment and Follow-up Phase
Time Frame: Up to Day 11 (Treatment Phase: at Day 4, Follow-up Phase: up to 7 days after the last dose)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21 | 21
Participants | 1 | 0

7. Secondary Outcome: Mean Seizure Frequency Per Day in Pretreatment Phase, Treatment Phase and Follow-up Phase
Description: Seizure frequency was based on number of seizures per day, calculated as the number of seizures over the entire time interval divided by the number of days in the interval.
Time Frame: Up to 39 days (Pretreatment Phase: up to 28 days; Treatment Phase: up to 4 days; Follow-up Phase: up to 7 days after the last dose)
Population: All participants who received at least 1 dose of study drug. Here "Number Analyzed" signifies participants who were evaluable for this outcome measure for POS and PGTC seizures.
Measure: Mean (Standard Deviation); unit: seizures per day
Arm/Group | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
Number analyzed (Participants) | 21 | 21 | 21
seizures per day
  POS | 0.46 (0.578) | 0.39 (0.838) | 0.24 (0.287)
  PGTC Seizures: number analyzed (Participants) | 1 | 1 | 1
  PGTC Seizures | 0 (NA) — Standard Deviation could not be estimated as only 1 participant was available for analysis. | 0 (NA) — Standard Deviation could not be estimated as only 1 participant was available for analysis. | 0 (NA) — Standard Deviation could not be estimated as only 1 participant was available for analysis.

8. Secondary Outcome: Plasma Concentration of Perampanel Before and After Switching From Oral Perampanel to 30-minute Intravenous Infusions of Perampanel
Time Frame: Pretreatment Phase-Day -1: Pre-dose, 0.5 hours, 1 hours and 1.5 hours post-dose; Treatment Phase-Day 1, Day 2, Day 3 and Day 4: Pre-dose and 0.5 hours after start of intravenous infusions
Population: All participants who received at least 1 dose of study drug. Here "Number Analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Pretreatment Phase: Oral Perampanel 8 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures received perampanel 8 mg (stable-dosage), tablets, orally, once daily for 28 days (Day -28 to Day -1) as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs. Eligible participants who completed Pretreatment Phase entered in Treatment Phase.
- Pretreatment Phase: Oral Perampanel 10 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures received perampanel 10 mg (stable-dosage), tablets, orally, once daily for 28 days (Day -28 to Day -1) as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs. Eligible participants who completed Pretreatment Phase entered in Treatment Phase.
- Pretreatment Phase: Oral Perampanel 12 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures received perampanel 12 mg (stable-dosage), tablets, orally, once daily for 28 days (Day -28 to Day -1) as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs. Eligible participants who completed Pretreatment Phase entered in Treatment Phase.
- Treatment Phase: Intravenous Perampanel 8 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures were hospitalized and received perampanel 8 mg (stable-dosage) equivalent to the oral dose, as intravenous infusion for 30 minutes, once daily on Day 1 to Day 4 as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs.
- Treatment Phase: Intravenous Perampanel 10 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures were hospitalized and received perampanel 10 mg (stable-dosage) equivalent to the oral dose, as intravenous infusion for 30 minutes, once daily on Day 1 to Day 4 as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs.
- Treatment Phase: Intravenous Perampanel 12 mg/Day: Participants with POS with or without secondarily generalized seizures or PGTC seizures were hospitalized and received perampanel 12 mg (stable-dosage) equivalent to the oral dose, as intravenous infusion for 30 minutes, once daily on Day 1 to Day 4 as an adjunctive therapy along with 1 to a maximum of 3 marketed concomitant AEDs.
Arm/Group | Pretreatment Phase: Oral Perampanel 8 mg/Day | Pretreatment Phase: Oral Perampanel 10 mg/Day | Pretreatment Phase: Oral Perampanel 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 mg/Day | Treatment Phase: Intravenous Perampanel 10 mg/Day | Treatment Phase: Intravenous Perampanel 12 mg/Day
Number analyzed (Participants) | 11 | 5 | 5 | 11 | 5 | 5
nanogram per milliliter (ng/mL)
  Day -1: Pre-dose: number analyzed (Participants) | 11 | 5 | 5 | 0 | 0 | 0
  Day -1: Pre-dose | 430 (336) | 352 (172) | 556 (255) |  |  |
  Day -1: 0.5 hour post-dose: number analyzed (Participants) | 11 | 5 | 5 | 0 | 0 | 0
  Day -1: 0.5 hour post-dose | 464 (369) | 435 (216) | 608 (271) |  |  |
  Day -1: 1 hour post-dose: number analyzed (Participants) | 11 | 5 | 5 | 0 | 0 | 0
  Day -1: 1 hour post-dose | 538 (385) | 499 (226) | 664 (282) |  |  |
  Day -1: 1.5 hour post-dose: number analyzed (Participants) | 11 | 5 | 5 | 0 | 0 | 0
  Day -1: 1.5 hour post-dose | 555 (356) | 521 (227) | 658 (284) |  |  |
  Day 1: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 5 | 5
  Day 1: Pre-dose |  |  |  | 402 (304) | 316 (156) | 554 (234)
  Day 1: 0.5 hour post-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 5 | 5
  Day 1: 0.5 hour post-dose |  |  |  | 609 (303) | 591 (172) | 837 (282)
  Day 2: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 4 | 5
  Day 2: Pre-dose |  |  |  | 382 (298) | 297 (170) | 540 (232)
  Day 2: 0.5 hour post-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 4 | 5
  Day 2: 0.5 hour post-dose |  |  |  | 614 (315) | 520 (184) | 760 (261)
  Day 3: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 4 | 5
  Day 3: Pre-dose |  |  |  | 372 (277) | 296 (175) | 560 (256)
  Day 3: 0.5 hour post-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 4 | 5
  Day 3: 0.5 hour post-dose |  |  |  | 557 (301) | 547 (169) | 815 (276)
  Day 4: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 4 | 5
  Day 4: Pre-dose |  |  |  | 394 (307) | 297 (184) | 552 (259)
  Day 4: 0.5 hour post-dose: number analyzed (Participants) | 0 | 0 | 0 | 11 | 4 | 5
  Day 4: 0.5 hour post-dose |  |  |  | 554 (300) | 541 (209) | 841 (312)

ADVERSE EVENTS:
Time Frame: Up to 60 days (Pretreatment Phase: up to 28 days, Treatment Phase: up to 4 days, Follow-up Phase: up to 28 days after the last dose)
Description: All participants who received at least 1 dose of study drug.
Arm/Group | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/21 | 2/21
Other Adverse Events (participants affected / at risk) | 2/21 | 11/21 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day (N=21) | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day (N=21) | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day (N=21)
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment Phase: Oral Perampanel 8 to 12 mg/Day (N=21) | Treatment Phase: Intravenous Perampanel 8 to 12 mg/Day (N=21) | Follow-up Phase: Oral Perampanel 8 to 12 mg/Day (N=21)
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Feeling abnormal (General disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 6 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03754582/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03754582/SAP_001.pdf